CLINICAL TRIAL: NCT01109953
Title: Improving Clinical PET/CT Image Quality in Retrospectively Reconstructed Breath-Hold Images
Status: Terminated | Type: Observational
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-054
Record Dates: First submitted 2010-04-20; First posted 2010-04-23 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer
Keywords: Lung; PET/CT scan; 10-054
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Breath-Hold PET/CT image: In addition to the standard clinical PET/CT images, we will provide a breath-hold PET/CT image set, using the same PET data for both.
  Interventions: Other: Breath-Hold PET/CT image set

INTERVENTIONS:
Other: Breath-Hold PET/CT image set — In addition to the standard clinical PET/CT images, we will provide a breath-hold PET/CT image set, using the same PET data for both. In order to spatially match PET, and therefore improve attenuation correction in the PET images, we will acquire a Breath-Hold CT at 310 mA over the same region covered by PET. The normal-organ doses accumulated from the additional 30 mA CT. The patient's breathing signal during CT and the whole body PET will be recorded using a video camera and in house developed software. We will compare the clinical PET/CT and Breath-Hold PET/CT in regards to lesion detection, lesion volume, and SUV quantification.

SUMMARY:
The patient has been referred for an FDG PET/CT scan. FDG is a form of sugar that contains a small amount of radioactivity; it is used to see the size and possible spread of cancer in the body.

Pictures of the body are taken on a machine called a PET/CT scanner. The purpose of this current study is to see if we, the investigators, can take clearer pictures of the tumor than we could with our routine scan method. This would allow us to better see how FDG is picked up by the tumor. PET/CT is presently one of the best tools for detecting cancer and determining its spread in the body. However, due to breathing motion, PET and CT images may become blurred and the location of the tumor on CT and PET images may not match. We have developed a new method that enables us to reduce image blurring and to measure the tumor more accurately on PET images. In this study we want to compare two kinds of images: those from the standard PET/CT scan, and the PET/CT scan pictures taken with our new method.

If successful, we may use this new method for clinical routine in the future.

ELIGIBILITY:
Inclusion Criteria:

* Participant is capable of providing written consent.
* 18 years of age or older.
* Patient with a known or suspected FDG-avid malignancy in the torso

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for whole body FDG PET/CT examination as part of their routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To determine if our breath-hold acquisition technique can be implemented in whole-body PET/CT scans. | at the time of scan
  Because PET events not satisfying the breathing amplitude selection criteria will be dropped off the final image set, it will be necessary to increase the acquisition time for the FOV's covering the thorax area from 3 min/bed to 5 min/bed to compensate for the reduction in statistics. This should result in a total increase of ~6 min for the whole body scan.

SECONDARY OUTCOMES:
To determine if whole body PET/CT improves spatial matching of PET and CT | at the time of scan
  to compare image quality, blurring, PET-to-CT mis-match, and lesion SUV of the standard PET images with the breath-hold ones.

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schoder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm